CLINICAL TRIAL: NCT04653766
Title: A Phase I, Double Blind, Placebo Controlled, Single Ascending Dose Study of Intravenously Administered Ir-CPI to Evaluate Pharmacokinetics, Pharmacodynamics, Safety and Tolerability in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ir-CPI in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioxodes S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: Clin_IrCPI_101; 2019-002305-22 (EudraCT Number)
Record Dates: First submitted 2020-10-29; First posted 2020-12-04 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Antithrombotic; Intrinsic coagulation pathway

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Ir-CPI - Dose 1 (Experimental): Participants received a single intravenous dose of 1.5 mg/kg of Ir-CPI during 6 hours
  Interventions: Drug: Ir-CPI - Dose 1
- Ir-CPI - Dose 2 (Experimental): Participants received a single intravenous dose of 3.0 mg/kg of Ir-CPI during 6 hours
  Interventions: Drug: Ir-CPI - Dose 2
- Ir-CPI - Dose 3 (Experimental): Participants received a single intravenous dose of 6.0 mg/kg of Ir-CPI during 6 hours
  Interventions: Drug: Ir-CPI - Dose 3
- Ir-CPI - Dose 4 (Experimental): Participants received a single intravenous dose of 9.0 mg/kg of Ir-CPI during 6 hours
  Interventions: Drug: Ir-CPI - Dose 4
- Placebo (Placebo Comparator): Participants received a single intravenous dose of placebo during 6 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ir-CPI - Dose 1 — 6 participants received a single intravenous dose of 1.5 mg/kg of Ir-CPI during 6 hours
  Arms: Ir-CPI - Dose 1
Drug: Ir-CPI - Dose 2 — 6 participants received a single intravenous dose of 3.0 mg/kg of Ir-CPI during 6 hours
  Arms: Ir-CPI - Dose 2
Drug: Ir-CPI - Dose 3 — 6 participants received a single intravenous dose of 6.0 mg/kg of Ir-CPI during 6 hours
  Arms: Ir-CPI - Dose 3
Drug: Ir-CPI - Dose 4 — 6 participants received a single intravenous dose of 9.0 mg/kg of Ir-CPI during 6 hours
  Arms: Ir-CPI - Dose 4
Drug: Placebo — For each dose group, 2 additional participants received a single intravenous dose of placebo during 6 hours (8 in total).
  Arms: Placebo

SUMMARY:
The purpose of this First-in-Human study is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of Ir-CPI, a novel dual inhibitor of FXIIa and FXIa, following IV administration of single ascending doses in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all of the following inclusion criteria before being allowed to enter the study:

1. Have given written informed consent approved by the relevant Ethics Committee (EC) governing the site, indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
2. Male participants between 18 and 55 years of age, inclusive at screening.
3. Otherwise healthy with no clinically significant abnormalities as determined by medical history, physical examination, blood chemistry assessments, haematological assessments, coagulation and urinalysis, measurement of vital signs, and ECG. Isolated out-of-range values judged by the PI (or designated physician) to be of no clinical significance can be allowed. This determination must be recorded in the participant's source documents.
4. Have a body weight in the range of 50 to 90 kg inclusive at screening. Have a body mass index (BMI) of 19 to 28 kg/m2 inclusive at screening.
5. Agree to abstain from alcohol intake 24 hours before administration of study drug, during the in-patient period of the study and 24 hours prior to all other ambulatory visits, up until and including the discharge visit.
6. Agree not to use prescription medications within 14 days prior to study drug administration and through the duration of the study, unless approved by the PI and Sponsor medical monitor.
7. Non-smokers or abstinence from tobacco or nicotine-containing products for at least 3 months prior to screening.
8. Agree not to use over-the-counter (OTC) medications [including decongestants, antihistamines, and herbal medication (including herbal tea and St. John's Wort)], within 14 days prior to study drug administration through the discharge visit, unless approved by the PI and Sponsor medical monitor. Occasional use of paracetamol at recommended doses is allowed. Special rules apply for aspirin, corticosteroids and nonsteroidal anti-inflammatory drugs (NSAIDS (see exclusion criteria 6-7-8-9)
9. Venous access (both arms) sufficient to allow blood sampling and study drug administration as per protocol.
10. Participants and their partners of childbearing potential [meaning who are not surgically sterile (tubal ligation/obstruction or removal of ovaries or uterus) or post-menopausal (absence of menstrual periods for at least 12 consecutive months)] must be willing to use 2 methods of contraception: - a highly effective method of birth control starting at screening. Highly effective methods of birth control are defined as those that result in a low failure rate (i.e. Pearl Index less than 1% per year) when used consistently and correctly, such as implants, rings, patches, injectable or combined oral contraceptives, intrauterine devices (IUDs), or sexual abstinence (periodic abstinence e.g. calendar, ovulation, symptothermal, postovulation methods, declaration of abstinence for the duration of the trial, and withdrawal are not acceptable methods of contraception) . - and a local barrier form of contraception. Acceptable barrier methods are either the participant's use of a condom or the partner's use of an occlusive cap or diaphragm, or spermicides. Participants will not donate sperm from the selection visit and up to 90 days after the infusion. In case of sterile or vasectomised participants, no contraception will be required for their partners of childbearing potential.
11. Willing/able to adhere to the study visit schedule and other requirements, prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

If any of the following exclusion criteria apply, the participant must not enter the study:

1. Currently have or have a history of any clinically significant medical illness or medical disorders the PI considers should exclude the participant, including (but not limited to) cardiovascular disease, neuromuscular, haematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease.
2. History of personal or familial bleeding disorders; including prolonged or unusual bleeding.
3. History of deficiency in factor XII (FXII) or haemophilia type A (FVII) or type B (FIX) or type C (FXI).
4. History of cerebral bleeding (e.g. after a car accident), stroke and cerebrovascular accident (CVA).
5. Anamnestic history of Lyme disease or tick-borne encephalitis.
6. Use of Acetylsalicylic-Acid (ASA)-containing OTC medications within 1 month prior to screening.
7. Chronic administration of NSAIDs, chronic use of corticosteroids within 1 month prior to screening.
8. Chronic administration of clopidogrel, ticlopidin, dipyridamole, Coumadin-like anticoagulants, new oral anticoagulant dabigatran, rivaroxaban, apixaban or edoxaban within 3 months prior to screening.
9. Administration of unfractionated heparin, low molecular weight heparin, fibrinolytic agents and anti-FXa within 3 months prior to screening.
10. Have an active acute or chronic infection or diagnosed latent infection.
11. Systolic blood pressure (SBP) greater than 150 or less than 90 mmHg, diastolic blood pressure (DBP) greater than 90 or less than 50 mmHg, and heart rate (HR) greater than 100 or less than 40 bpm.
12. Acute clinically relevant illness within 7 days prior to study drug administration or have had a major illness or hospitalisation within 1 month prior to study drug administration.
13. Major or traumatic surgery within 12 weeks of screening.
14. Any participant who plans to undergo elective surgery within 4 weeks prior to study drug administration and through the discharge visit.
15. Positive serology test for HIV antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies at screening.
16. Recent history (within previous 6 months) of alcohol or drug abuse.
17. Have positive urine toxicology screen at screening or D -1 for substances of abuse including amphetamines, benzodiazepine, cocaine, opiates, barbiturate and cannabinoids.
18. Have a positive alcohol breath test at screening or D-1.
19. Consumes, on average, more than approximately 500 mg/day of caffeine (as contained in 5 cups of tea or coffee or 8 cans of caffeine-containing soda or other caffeinated products per day).
20. Donated blood (i.e. 500 mL) within 3 months before D1.
21. Have a history of active drug and/or food allergy or other active allergic disease requiring the constant use of medications, or a history of severe allergic reaction, angioedema or anaphylaxis.
22. Received any other experimental therapy or new investigational drug within 30 days or 5 half-lives (whichever is longer) of study drug administration.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-07-18 (Actual); Study Completion 2023-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- A.T.C. Pharma, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4 | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (12.2) | 35.2 (11.8) | 27.3 (7.6) | 34.8 (10.0) | 35.8 (11.4) | 33.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 8 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 8 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 6 | 6 | 6 | 6 | 8 | 32
Height [Mean (Standard Deviation); unit: cm] | 178.8 (4.4) | 175.3 (4.5) | 177.2 (4.9) | 174.8 (6.8) | 179.5 (6.9) | 177.3 (5.7)
Weight [Mean (Standard Deviation); unit: kg] | 78.43 (4.28) | 76.22 (9.24) | 77.25 (6.34) | 66.80 (7.93) | 72.96 (6.99) | 74.25 (7.84)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 24.52 (0.95) | 24.75 (2.47) | 24.65 (2.32) | 21.81 (1.63) | 22.68 (2.23) | 23.62 (2.24)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of the Safety Lab Parameter Activated Partial Thromboplastin Time (aPTT)
Description: These safety aPTT results were readily available to the PI for safety follow-up during and after the study drug administration. Safety aPTT was followed up "at the bedside" at regular time-points (as opposed to the PD biomarker aPTT, which was assessed by the central laboratory alongside the PK time-points). An aPTT ratio was calculated by dividing the aPTT value (in sec) of the specific time-point (aPTTt) by the baseline aPTT value (in sec) (aPTTbaseline) of the same participant (aPTT ratio = aPTTt/aPTTbaseline). The baseline time-point was considered as having an aPTT ratio of 1.
  Concerning the row titles, for example, Day 1 H02:00 corresponds to aPTT ratio results obtained on Day 1, 2 hours after the start of the infusion.
Time Frame: At pre-dose (baseline), 2, 4, 6, 8, 12, 24, 48, 72 hours post-dose and at the discharge visit (Day 10 ± 2 days)
Measure: Mean (Standard Deviation); unit: aPTT ratio
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
aPTT ratio
  Day 1 H00:00 (baseline) | 1.000 (0.000) | 1.000 (0.000) | 1.000 (0.000) | 1.000 (0.000) | 1.000 (0.000)
  Day 1 H02:00 | 1.600 (0.080) | 1.978 (0.068) | 2.405 (0.214) | 2.627 (0.126) | 0.986 (0.088)
  Day 1 H04:00 | 1.768 (0.123) | 2.262 (0.085) | 2.628 (0.260) | 2.875 (0.129) | 0.981 (0.077)
  Day 1 H06:00 | 1.860 (0.103) | 2.313 (0.060) | 2.775 (0.269) | 2.993 (0.196) | 0.994 (0.086)
  Day 1 H08:00 | 1.520 (0.100) | 1.832 (0.072) | 2.135 (0.208) | 2.367 (0.096) | 0.960 (0.091)
  Day 1 H12:00 | 1.308 (0.070) | 1.600 (0.102) | 1.848 (0.075) | 2.077 (0.046) | 0.970 (0.075)
  Day 2 H24:00 | 1.162 (0.056) | 1.352 (0.122) | 1.627 (0.114) | 1.725 (0.056) | 0.973 (0.077)
  Day 3 H48:00 | 1.033 (0.041) | 1.123 (0.132) | 1.313 (0.063) | 1.377 (0.064) | 0.983 (0.108)
  Day 4 H72:00 | 1.020 (0.036) | 1.083 (0.056) | 1.143 (0.067) | 1.182 (0.046) | 0.974 (0.071)
  Day 10 (discharge visit) | 1.003 (0.029) | 1.017 (0.072) | 1.027 (0.046) | 0.993 (0.043) | 0.993 (0.093)

2. Secondary Outcome: Measurement of the Maximum Plasma Concentration (Cmax) of Ir-CPI
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 6.5, 7, 7.5, 8, 10, 12, 16, 24, 48, 72, 96, 144 hours (144 hours for Dose 4 only)
Population: Pharmacokinetic set (PKS): all of the included participants who were administered a complete infusion of study drug without major protocol deviation affecting PK evaluation.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 958.8 (98.6) | 2013.2 (228.2) | 3752.5 (422.3) | 6288.3 (757)

3. Secondary Outcome: Measurement of the Time to Reach Maximum Plasma Concentration (Tmax) of Ir-CPI
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 6.5, 7, 7.5, 8, 10, 12, 16, 24, 48, 72, 96, 144 hours (144 hours for Dose 4 only)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 6 (0) | 6 (0) | 6 (0) | 6 (0)

4. Secondary Outcome: Measurement of the Area Under the Plasma Concentration-time Curve From Time Zero to 6h (AUC0-6) and From Time Zero to Time of Infinity (AUCinf)
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 6.5, 7, 7.5, 8, 10, 12, 16, 24, 48, 72, 96, 144 hours (144 hours for Dose 4 only)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/mL
  AUC0-6h | 3648.0 (250.7) | 7915.5 (1210.2) | 15184.7 (1863.9) | 24683.2 (5069.5)
  AUC0-inf | 13446.3 (1208.2) | 26573.3 (2037.3) | 53541.5 (3832.6) | 104509.8 (10124.8)

5. Secondary Outcome: Measurement of the Effect of Ir-CPI on the Activated Partial Thromboplastin Time (aPTT)
Description: The activated partial thromboplastin time (aPTT) is used as a pharmacodynamic marker. No data were available for the Ir-CPI 1.5 mg/kg group because the results were not usable due to plasma preparation and method repeatability problems. An aPTT ratio was calculated by dividing the aPTT value (in sec) of the specific time-point (aPTTt) by the baseline aPTT value (in sec) (aPTTbaseline) of the same participant (aPTT ratio = aPTTt/aPTTbaseline). The baseline time-point (Day 1 H00:00) was considered as having an aPTT ratio of 1.
  Concerning the row titles, for example, Day 1 H02:00 corresponds to aPTT ratio results obtained on Day 1, 2 hours after the start of the infusion.
Time Frame: Pre-dose (baseline), 0.5, 1, 1.5, 2, 4, 6, 6.5, 7, 7.5, 8, 10, 12, 16, 24, 48, 72, 96 hours post-dose and at the discharge visit (Day 10 ± 2 days)
Population: This analysis was performed on the Pharmacodyamic Set (PDS): all of the included participants who completed the study without any protocol deviation affecting PD evaluation and with at least one available post-baseline PD data point.
Measure: Mean (Standard Deviation); unit: aPTT ratio
Arm/Group | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 8
aPTT ratio
  Day 1 H00:00 (baseline) | 1.000 (0.000) | 1.000 (0.000) | 1.000 (0.000) | 1.000 (0.000)
  Day 1 H00:30 | 1.535 (0.093) | 1.825 (0.133) | 2.218 (0.358) | 0.982 (0.115)
  Day 1 H01:00 | 1.707 (0.073) | 2.085 (0.131) | 2.397 (0.296) | 0.962 (0.097)
  Day 1 H01:30 | 1.827 (0.091) | 2.225 (0.122) | 2.533 (0.185) | 0.982 (0.102)
  Day 1 H02:00 | 1.915 (0.079) | 2.367 (0.143) | 2.692 (0.214) | 0.972 (0.094)
  Day 1 H04:00 | 2.148 (0.141) | 2.583 (0.218) | 2.822 (0.096) | 0.970 (0.094)
  Day 1 H06:00 | 2.207 (0.119) | 2.652 (0.260) | 3.050 (0.189) | 0.973 (0.116)
  Day 1 H06:30 | 2.045 (0.109) | 2.442 (0.222) | 2.798 (0.184) | 0.982 (0.109)
  Day 1 H07:00 | 1.917 (0.105) | 2.240 (0.154) | 2.558 (0.113) | 0.972 (0.101)
  Day 1 H07:30 | 1.842 (0.093) | 2.103 (0.131) | 2.402 (0.206) | 0.950 (0.121)
  Day 1 H08:00 | 1.775 (0.097) | 2.098 (0.161) | 1.098 (0.161) | 0.945 (0.102)
  Day 1 H10:00 | 1.638 (0.113) | 1.942 (0.154) | 2.230 (0.108) | 0.922 (0.117)
  Day 1 H12:00 | 1.540 (0.120) | 1.842 (0.119) | 2.137 (0.116) | 0.952 (0.106)
  Day 1 H16:00 | 1.428 (0.115) | 1.705 (0.102) | 1.947 (0.096) | 0.987 (0.075)
  Day 2 H24:00 | 1.312 (0.151) | 1.585 (0.107) | 1.718 (0.116) | 0.965 (0.103)
  Day 3 H48:00 | 1.125 (0.109) | 1.277 (0.106) | 1.390 (0.064) | 0.945 (0.117)
  Day 4 H72:00 | 1.025 (0.107) | 1.113 (0.118) | 1.172 (0.053) | 0.988 (0.133)
  Day 5 H96:00 | 0.990 (0.094) | 1.037 (0.088) | 1.062 (0.049) | 0.942 (0.098)
  Day 10 (discharge visit) | 0.972 (0.078) | 0.967 (0.072) | 0.978 (0.067) | 0.985 (0.128)

6. Secondary Outcome: Measurement of the Effect of Ir-CPI on Factor XI Activity
Description: The method is a clotting assay where all the clotting factors are present (constant and in excess, brought by the deficient plasma), excepted for FXI, which is brought by the diluted tested plasma, and clotting is triggered with cephalin, activator and calcium (aPTT). FXI is the limiting factor and clotting time is inversely proportional to the concentration of FXI. There is an inverse linear relationship between the percentage of FXI activity and the corresponding clotting time. Central laboratory normal ranges for Factor XI activity are between 65 and 150 %.
  Concerning the row titles, for example, Day 1 H02:00 corresponds to the percentage of FXI activity obtained on Day 1, 2 hours after the start of the infusion.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of Factor XI activity
Groups:
- Ir-CPI - Dose 2: Participants received a single intravenous dose of 3.0 mg/kg or Ir-CPI during 6 hours
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Percentage of Factor XI activity
  Day 1 H00:00 (baseline) | 112.3 (23.9) | 103.7 (22.2) | 89.2 (9.8) | 94.5 (8.4) | 95.9 (12.4)
  Day 1 H00:30 | 98.7 (20.1) | 85.5 (15.6) | 61.8 (8.3) | 58.8 (8.1) | 99.5 (10.2)
  Day 1 H01:00 | 94.8 (23.4) | 79.5 (14.3) | 53.3 (7.1) | 54.7 (7.6) | 104.8 (12.2)
  Day 1 H01:30 | 98.0 (18.2) | 73.3 (11.3) | 49.8 (6.3) | 50.0 (7.6) | 99.3 (14.2)
  Day 1 H02:00 | 91.5 (19.1) | 70.8 (12.8) | 46.2 (6.0) | 47.2 (7.2) | 100.1 (10.8)
  Day 1 H04:00 | 88.8 (19.1) | 64.0 (10.8) | 42.5 (5.5) | 41.7 (4.1) | 106.6 (13.8)
  Day 1 H06:00 | 85.5 (16.5) | 61.7 (12.3) | 41.3 (3.3) | 40.5 (5.5) | 106.6 (12.7)
  Day 1 H06:30 | 88.7 (19.5) | 67.7 (10.8) | 49.5 (6.7) | 45.3 (7.0) | 104.9 (13.0)
  Day 1 H07:00 | 91.3 (25.9) | 70.7 (13.9) | 49.2 (4.4) | 47.0 (8.4) | 101.6 (10.9)
  Day 1 H07:30 | 91.7 (23.9) | 74.5 (11.7) | 51.0 (5.6) | 47.8 (8.0) | 100.5 (14.5)
  Day 1 H08:00 | 92.8 (20.8) | 73.8 (12.0) | 54.8 (4.3) | 50.7 (9.1) | 106.4 (15.4)
  Day 1 H10:00 | 99.3 (28.1) | 83.2 (14.5) | 61.0 (6.9) | 56.7 (11.2) | 106.4 (14.9)
  Day 1 H12:00 | 102.7 (25.0) | 87.0 (16.1) | 61.5 (7.1) | 59.5 (9.7) | 101.0 (11.5)
  Day 1 H16:00 | 101.8 (25.7) | 89.0 (15.2) | 65.3 (8.0) | 63.5 (11.0) | 98.4 (11.1)
  Day 2 H24:00 | 116.0 (35.8) | 92.7 (15.8) | 73.2 (9.9) | 71.2 (11.3) | 104.8 (8.5)
  Day 3 H48:00 | 117.8 (21.9) | 104.7 (24.8) | 85.8 (13.8) | 81.5 (12.7) | 104.0 (9.5)
  Day 4 H72:00 | 136.8 (81.0) | 104.5 (20.9) | 92.8 (6.9) | 86.7 (17.3) | 105.5 (7.8)
  Day 5 H96:00 | 110.8 (23.0) | 105.5 (24.2) | 90.0 (11.0) | 97.2 (19.1) | 107.4 (14.0)
  Day 10 (discharge visit) | 111.3 (28.6) | 107.7 (17.9) | 93.2 (9.3) | 99.3 (16.8) | 103.4 (11.7)

7. Secondary Outcome: Measurement of the Effect of Ir-CPI on Factor XII Activity
Description: The method is a clotting assay where all the clotting factors are present (constant and in excess, brought by the deficient plasma), excepted for FXII, which is brought by the diluted tested plasma, and clotting is triggered with cephalin, activator and calcium (aPTT). FXII is the limiting factor and clotting time is inversely proportional to the concentration of FXII. There is an inverse linear relationship between the percentage of FXII activity and the corresponding clotting time. Central laboratory normal ranges for Factor XII activity are between 50 and 150 %.
  Concerning the row titles, for example, Day 1 H02:00 corresponds to the percentage of FXII activity obtained on Day 1, 2 hours after the start of the infusion.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of Factor XII activity
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Percentage of Factor XII activity
  Day 1 H00:00 (baseline) | 105.0 (24.9) | 94.8 (20.8) | 101.5 (36.9) | 100.0 (15.9) | 111.0 (28.3)
  Day 1 H00:30 | 93.0 (12.8) | 68.8 (18.7) | 60.8 (26.1) | 42.3 (9.7) | 114.0 (29.6)
  Day 1 H01:00 | 83.5 (21.2) | 62.2 (17.7) | 45.8 (21.7) | 35.0 (5.3) | 119.1 (20.4)
  Day 1 H01:30 | 82.7 (23.6) | 53.3 (15.0) | 43.8 (22.6) | 29.3 (5.3) | 111.4 (25.6)
  Day 1 H02:00 | 76.0 (16.3) | 49.3 (12.5) | 32.7 (13.7) | 26.3 (5.0) | 113.5 (26.7)
  Day 1 H04:00 | 68.5 (16.4) | 40.5 (10.6) | 27.5 (12.8) | 24.8 (4.6) | 117.0 (29.1)
  Day 1 H06:00 | 64.8 (12.8) | 38.2 (5.7) | 26.7 (11.9) | 24.2 (7.4) | 116.4 (26.3)
  Day 1 H06:30 | 69.5 (16.8) | 45.8 (11.8) | 33.3 (13.6) | 25.8 (5.9) | 116.3 (25.2)
  Day 1 H07:00 | 75.0 (21.1) | 47.0 (11.0) | 35.8 (14.7) | 29.8 (8.2) | 116.8 (29.2)
  Day 1 H07:30 | 75.2 (18.2) | 53.3 (14.4) | 39.0 (17.1) | 31.2 (8.1) | 115.9 (25.5)
  Day 1 H08:00 | 77.7 (20.2) | 54.7 (12.1) | 44.3 (18.3) | 34.0 (7.6) | 117.4 (26.7)
  Day 1 H10:00 | 90.3 (22.9) | 65.5 (15.7) | 54.2 (21.7) | 40.5 (8.8) | 118.3 (24.3)
  Day 1 H12:00 | 91.3 (21.6) | 71.3 (14.5) | 58.5 (23.8) | 42.3 (9.7) | 113.6 (27.4)
  Day 1 H16:00 | 89.7 (23.0) | 73.8 (18.6) | 61.0 (24.2) | 49.8 (11.7) | 112.8 (29.0)
  Day 2 H24:00 | 104.8 (25.9) | 80.3 (16.4) | 78.8 (31.3) | 59.3 (14.6) | 116.5 (27.0)
  Day 3 H48:00 | 128.7 (27.6) | 96.7 (15.4) | 92.0 (35.8) | 79.7 (21.0) | 118.1 (28.6)
  Day 4 H72:00 | 121.5 (29.2) | 98.3 (15.9) | 112.0 (13.3) | 89.5 (24.2) | 120.4 (29.6)
  Day 5 H96:00 | 123.5 (27.3) | 100.5 (17.4) | 102.5 (36.5) | 100.2 (23.8) | 121.6 (29.3)
  Day 10 (discharge visit) | 122.0 (26.9) | 102.2 (20.2) | 104.0 (35.3) | 107.2 (23.8) | 114.3 (27.5)

ADVERSE EVENTS:
Time Frame: From screening visit through last extra-ambulatory visit [Day 90 or Day 180 (in case of anti-drug antibodies at Day 90)]
Arm/Group | Ir-CPI - Dose 1 | Ir-CPI - Dose 2 | Ir-CPI - Dose 3 | Ir-CPI - Dose 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 1/6 | 0/8
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 5/6 | 6/6 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ir-CPI - Dose 1 (N=6) | Ir-CPI - Dose 2 (N=6) | Ir-CPI - Dose 3 (N=6) | Ir-CPI - Dose 4 (N=6) | Placebo (N=8)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyarthritis acute (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ir-CPI - Dose 1 (N=6) | Ir-CPI - Dose 2 (N=6) | Ir-CPI - Dose 3 (N=6) | Ir-CPI - Dose 4 (N=6) | Placebo (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (3) | 1 (2) | 3 (3) | 1 (2)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (7) | 3 (6) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sebaceous cyst excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT04653766/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04653766/SAP_001.pdf